CLINICAL TRIAL: NCT01151176
Title: Phase IV Study of a Feasible Insulin Algorithm for Glycemic Control in Patients With Acute Coronary Syndrome
Brief Title: Feasible Insulin Algorithm for Glycemic Control in Patients With Acute Coronary Syndrome
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative problems makes changes in hospital staff New clinical research team will restart
Sponsor: Universidade Positivo (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Silmara A O Leite, PhD, Universidade Positivo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-001
Record Dates: First submitted 2010-03-04; First posted 2010-06-28 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Intensive Insulin Therapy; Glucose control; Acute Coronary Syndrome; Intensive Care
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Active Comparator): Intensive Insulin Therapy
  Interventions: Drug: Regular Insulin
- Regular Insulin (Other): Sub Cutaneous Regular Insulin
  Interventions: Drug: Regular Insulin

INTERVENTIONS:
Drug: Regular Insulin — 1,8U Regular insulin/h from 180mg/dL of blood glucose increasing each hour according to capillary blood glucose. Between 100-150mg/dL keep infusion and bellow 100mg/dL stop infusion
  Other Names: Novolin R
  Arms: Insulin
Drug: Regular Insulin — Regular Insulin SC according to Blood Glucose(mg/dL) and Insulin Sensitive with usual dose describe and less 2U for sensitive and plus 2U for insulin resistant:
  Blood Glucose >141-180=4U ;181-220=6U; 221-260=8U; 261-300=10U;301-350=12U; 351-400=14U; > 400=16U
  Other Names: Novolin R
  Arms: Regular Insulin

SUMMARY:
The study aims to demonstrate that a simple intravenous insulin algorithm can be implemented in Latin America and will result in safe and better glucose control in patients with Acute Coronary Syndrome (ACS) compared with SC insulin.

DETAILED DESCRIPTION:
The proposed study is a one center open-label randomized controlled clinical trial.Coronary Intensive Care of one hospital in the city of Curitiba, PR, Brazil will be assessed.

Consenting eligible subjects will be randomized to either the intensive insulin infusion therapy group (ITG) or the conventional therapy group (CTG).

This particular insulin infusion was adapted of a protocol has been used before in patients who underwent to cardiothoracic surgery and its efficacy has been reported in the literature.

The control group will be selected following the same set of inclusion and exclusion criteria. Patients will be randomized to receive SC regular insulin 4 times daily (before meals and bedtime) or every 6 hours if they are NPO .

Data will be collected for history of diabetes, heart disease ; hypertension; hyperlipidemia; Current smoker; Cardiac treatment (Aspirin, Beta Blockers, ACE inhibitor/A2RB, Nitrates, Statin, Fibrate) Diabetes treatment(Insulin, Metformin, Sulphonylureas) Data will be collect for Baseline BGL , A1C level, Troponin, CPK, CKP-Mb, K, Creatinine. Classify Infarct type : Anterior/anteroseptal, Inferior, Non-ST-segment elevation myocardial infarction, Not classified Cardiac intervention : PTCA , Thrombolysis,No reperfusion, Heparin or low-molecular weight heparin.

Subjects allocated to ITG will be placed on Grady Health System protocol, and those in CTG will follow the sliding scale nomograms. Insulin replacement will start during first 24h of admission. Patients will be followed during all hospital stay, but only at ICU the CIII and SC insulin replacement will be compared. After ICU discharge they will follow they will be followed by their physician with recommendations to keep blod glucose<180mg/dL.

Patients will be followed up to 90 days after hospital discharge with phone call.Subjects will be contacted to obtain information regarding the occurrence of cardiovascular events following discharge. If the subject is not contactable, the next of kin and/or the subject's general practitioner would be contacted. Where no information could be obtained, a request will be made to the Department of Births and Deaths.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 or older
* Evidence of AMI within the last 24 h (troponin-T >0.1mcg/l) or electrographic criteria of ST-segment elevation in two limb leads)
* Evidence of Unstable Angina
* Blood glucose >180mg/dL at admission with or without preexisting diabetes
* Willing to give informed consent
* Access to telephone communications after hospital discharge

Exclusion Criteria:

* Under 18 years of age
* Pregnant or lactating female
* Diabetes ketoacidosis
* Heart failure
* Cardiogenic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Differences in daily blood glucose mean concentration between treatment groups | 18 months

SECONDARY OUTCOMES:
Evaluating the performance of the insulin drip protocol to maintain target glucose control(TGC) | 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Silmara AO Leite, PhD, MD, Principal Investigator — Universidade Positivo; Guilhermo E Umpierrez, MD, Study Chair — Emory University
Locations (2):
- Emory University School of Medicine, Atlanta, Georgia, United States
- Hospital Cruz Vermelha Brasileira-Filial do Estado do Paraná, Curitiba, Paraná, Brazil